CLINICAL TRIAL: NCT03272503
Title: A Phase II Randomized, Placebo-Controlled, Double Blinded, Multi-Centre Clinical Trial of Pimozide in Patients With Amyotrophic Lateral Sclerosis
Brief Title: A Clinical Trial of Pimozide in Patients With Amyotrophic Lateral Sclerosis (ALS)
Acronym: Pimozide2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: ALS Canada (Unknown); Brain Canada (Other)
Responsible Party: Principal Investigator, DR. LAWRENCE KORNGUT, M.D. Director Calgary ALS and Motor Neuron Disease Clinic, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pimozide2_ALS-002
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: ALS; Amyotrophic Lateral Sclerosis
Keywords: Pimozide
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Pimozide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 Pimozide 2 mg (current) or 4 mg/day (study initiation) (Experimental): Pimozide will be initiated at 2 mg once daily. The maximum dose will then be administered for a target period of 22 weeks.
  Interventions: Drug: Pimozide 2mg/day (current) or 4 mg/day (study initiation)
- Group 2 Placebo (Placebo Comparator): Placebo tablets will be utilized and administered in an identical manner for subjects in Group 1
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Pimozide 2mg/day (current) or 4 mg/day (study initiation) — Pimozide 2mg tablets will be taken once daily.
  Arms: Group 1 Pimozide 2 mg (current) or 4 mg/day (study initiation)
Drug: Placebo Oral Tablet — Identical matching placebo lactose tablets
  Arms: Group 2 Placebo

SUMMARY:
This study will look at whether Pimozide may help to slow the progression of Amyotrophic Lateral Sclerosis.

100 people from several Canadian centres with ALS who have provided their consent will be randomly assigned into one of 2 groups. The first group will receive a dose of up to 2mg of Pimozide per day and the second group will receive placebo (lactose tablets). Subjects will be assigned randomly (like by a flip of a coin) to receive either Pimozide 2 mg per day or placebo tablets. There will be a fifty-fifty chance of receiving Pimozide or placebo.

Participants will be on study medication up to 22 weeks, and on study up to 26 weeks. There are 8 clinic visits and 1 phone visit over the course of the Treatment Phase of the study. The second phase which is Observational, is optional with follow-up for up to 5 years from the end of the Treatment Phase.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) or Lou Gehrig's disease is a neuromuscular disease that results in rapid decline in normal muscle function and tone leading to difficulties with mobility, eating, drinking, breathing, sleeping, and communicating. The disease is progressive and no cure currently exists. Most people diagnosed with ALS succumb within 3 to 5 years. Rilutek® (riluzole) has been approved as a treatment to slow progression of ALS, but is minimally effective with mean increase in survival of only a few months. Radicava® or Radicut® (edaravone) has recently been approved in Canada, USA, Japan and South Korea.

Muscular dysfunction present in people with ALS is caused by nerve breakdown and a dysfunction in the communication between the muscles and the nerves. The area where these communications occur is called the neuromuscular junction. Some recent studies have focused on using different medications to enhance communication at the neuromuscular junction with the goal of improving muscle function as a result. This approach is unproven but may help to slow the progression of the disease.

Pimozide is a medication that has been demonstrated to enhance communication at the neuromuscular junction in fish and mice. This study will look at whether Pimozide may help to slow the progression of ALS.

There are two parts to this study.

Treatment Phase: In the first part of this study, 100 people from several Canadian centres with ALS who have provided their consent will be randomly assigned into one of 2 groups. The first group will receive a dose of up to 2mg of Pimozide per day and the second group will receive placebo (lactose tablets). Subjects will be assigned randomly (like by a flip of a coin) to receive either Pimozide 2 mg per day or placebo tablets. There will be a fifty-fifty chance of receiving Pimozide or placebo.

Each Pimozide tablet contains 2 mg of Pimozide. The matching placebo tablets for this study will look exactly like the Pimozide tablets. Placebos are used in clinical trials to find out if the results observed in the study are due the drug being tested, or for other reasons.

Neither the subject nor their doctor will know which group a patient belongs to. However, if an emergency should arise, information about a treatment group will be shared with their doctor to ensure appropriate medical care. Participants will take their treatment once a day, every day for about 22 weeks. The total time in the study from the screen visit up until the last phone call communication is about 26 weeks.

Observational Phase: The second part of this study is optional. It is each subject's decision whether to participate only in the first part of this study, or in both parts of the study, or not at all. In the second part of this study, the Canadian Neuromuscular Disease Registry (CNDR) will collect data on overall ALS progression using the Revised ALS Functional Rating Scale (ALSFRS-R) and breathing using Vital Capacity data collected during breathing tests. This information will be collected from a subject medical record following each routine clinical appointment. Data will be collected at each routine clinic visit for up to 5 years from the end of the first part of the study. There will be no extra visits for this part of the study beyond routine ALS clinic visits.

The information collected during this part of the study will be used to compare the progression of ALS, after the clinical trial is completed, among the two treatment types (Placebo or 2 mg per day). By analyzing this information, the researchers conducting this study hope to determine if Pimozide may help to slow the progression of ALS. To participate in this part of the study consent must be provided to join the CNDR. A subject who hasn't already provided their CNDR consent, and wishes to participate in this part of the study will be given a CNDR consent form to review and sign in addition to this consent form. A subject already participating in the CNDR will just need to sign the main study consent form.

ELIGIBILITY:
Inclusion Criteria:

1. Patients classified as having clinically definite, clinically probable, clinically probable (laboratory-supported) or clinically possible ALS according to the El-Escorial diagnostic criteria for ALS (see Appendix 2).
2. Able to comprehend and willing to sign Informed Consent Form (ICF).
3. Age 18 years of age or greater.
4. ALS Symptom onset of muscle weakness or speech impairment no more than 48 months prior to screen visit. Fasiculations should not be considered.
5. Slow Vital Capacity (SVC) greater than or equal to 50% predicted for sex, age and height at screen.
6. Has the ability to swallow tablets/capsules whole at study entry.
7. Subject with clinical laboratory findings within the normal range or, if outside the normal range, determined by the Investigator at the Screening visit to be not clinically significant.
8. If the subject is taking Riluzole the dose must be stable for 30 days prior to the randomization visit. Riluzole cannot be initiated during the study.
9. If the subject is receiving Edaravone therapy, the dose must be stable for at least 1 cycle of infusion treatments before the randomization visit.

Exclusion Criteria:

1. History of laryngeal spasm, dystonia, or akathisia.
2. Diagnosis of ongoing symptomatic Restless Leg Syndrome or undergoing current treatment for Restless Leg Syndrome. If subject has symptoms that resemble or have the potential to be Restless Leg Syndrome, then further investigation should be undertaken to confirm or rule out diagnosis of Restless Leg Syndrome.
3. Any history of moderate or severe traumatic brain injury as defined by a Glasgow Coma Scale Score of less than 13/15 at any time point following a head injury without sedation or other reason for a decreased level of consciousness.
4. History of neuroleptic malignant syndrome.
5. History of hypersensitivity or serious adverse reaction(s) to a neuroleptic medication.
6. History of hyponatremia < 130 mmol/L
7. Subject with aspartate aminotransferase (AST) or alanine aminotransferase (ALT) value >3.0 times the upper limit of normal at the Screening visit.
8. Current heparin or warfarin use.
9. History of hepatic and/or renal impairment that may affect pimozide metabolism
10. History of current pregnancy, or breastfeeding women, or women planning to become pregnant. Female subjects of childbearing potential (sexually mature female who has not undergone a hysterectomy or who has not been post-menopausal for 12 consecutive months), must practise effective contraception during the study and be willing and able to continue contraception until the Follow-up phone visit after discontinuing study medication. Abstinence can be considered an acceptable method of contraception at the discretion of the investigator.
11. Current antipsychotic use
12. Presence of central nervous system depression, comatose states, liver disorders, renal insufficiency, and blood dyscrasias
13. Presence of Parkinson's syndrome
14. Presence of major depressive disorders as determined by site Investigator.
15. History of clinically significant ECG abnormalities at screen visit, including QTc>500ms.
16. History of congenital long QT syndrome or with a family history of this syndrome and in patients with a history of cardiac arrhythmias or Torsade de Pointes.
17. Presence of acquired long QT interval, and/or concomitant use of drugs known to prolong the QT interval (TCAs, opioids such as methodone, quinolone antibiotics (ciprofloxacin), antimalarials (quinine), Detrol, azole antifungals, Class 1A, III and 1C antiarrhythmics, and macrolide antibiotics.
18. Presence of clinically significant bradycardia (heart rate < 50 beats per minute)
19. Presence of hypokalemia or hypomagnesemia.
20. The concomitant use of CYP 3A4-inhibiting drugs such as azole antimycotics, antiviral protease inhibitors, macrolide antibiotics and nefazodone.
21. The concomitant use of CYP 2D6-inhibiting drugs such as quinidine is also contraindicated.
22. Concomitant use of serotonin reuptake inhibitors, such as, sertraline, paroxetine, citalopram and escitalopram.*
23. Has taken any compound under current or known future study as a potential therapy (including Withania) for ALS less than 30 days prior to dosing OR history of exposure to stem cell therapy for treatment of ALS at any time.
24. Current Neurological impairment due to a condition other than ALS:

    1. Subject in whom causes of neuromuscular weakness other than ALS have not been excluded.
    2. Subject with a diagnosis of other neurodegenerative diseases (e.g., Parkinson's disease, Frontotemporal dementia, Alzheimer's disease, etc.)
25. Use of non-invasive ventilation (BiPAP or CPAP) prior to Baseline visit at any time.
26. Cognitive impairment as determined by the Site Investigator, subject must not have an impaired ability to provide informed consent and must be able to understand study processes and comply with study procedures.
27. Extrapyramidal Symptom Rating Scale (ESRS) Parkinsonism score of 2 on 2 items or a score > 3 on 1 item; OR Dystonia score of >3 on at least 1 item or a score of 2 on 2 items; OR Tardive Dyskinesia score of >3 on at least 1 item or a score of 2 on 2 items. Do not consider scores greater than 3 for Tremor in any region if due to Benign Essential, Exaggerated, or Physiological Tremor.
28. The concomitant use of SSRIs and tricyclic antidepressants (e.g. amitriptyline, amoxaprine, desipramine, doxepin, imipramine, nortriptyline, protripyline, trimipramine) - and Tolterodine (Detrol) CYP2D6 inhibitor.

    * Prohibited medications such as tricyclic antidepressants, antimalarials, and serotonin reuptake inhibitors,(ie sertraline, paroxetine, citalopram, fluoxetine, vilazodone and escitalopram) may be weaned to full discontinuation at the screening visit after consent has been signed (no study procedures including adjustments to medication may occur until informed consent has been provided).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-10-27 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in ALS Functional Rating Scale-Revised (ALSFRS-R) | Change from Baseline (week 2), at visit each of visit weeks 4, 8,12,16,20, week 24 Final Study visit, and week 26 follow-up phone call. Will also be done for a study drug withdrawal visit or if applicable, an edaravone initiation visit.
  The Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised (ALSFRS-R) consists of a 12 item questionnaire which asks about function in certain daily activities. Takes around 5-10 mins with a study staff member.

SECONDARY OUTCOMES:
Change in Slow Vital Capacity (SVC) | Change from screen, at each of visit weeks 8, week 16, and week 24 Final Study visit. Will also be done for a study drug withdrawal visit or if applicable, an edaravone initiation visit.
  The SVC is the maximum volume of air which can be exhaled after a deep breath in, during a slow/steady maneuver. A nose clip will be placed on the nose during the testing.
Change in Decremental responses on repetitive nerve stimulation (DRRNS) | Change from Baseline (week 2) at week 24 Final Study visit. Will also be done for a study drug withdrawal visit or if applicable, an edaravone initiation visit.
  Repetitive Nerve Stimulation is where electrical stimulation is applied to a motor nerve repeatedly several times per second. This will involve testing each thumb.
Change in Motor Power - the MRC (Medical Research Council) Sum Score | Change from screen, at each of week 8, week 16, and week 24 Final Study visit. Will also be done for a study drug withdrawal visit or if applicable, an edaravone initiation visit.
  Assessment of Muscle Strength
Change in Common Terminology Criteria for Adverse Events (CTCAE) will be entered for each visit for adverse effect profile analysis | Change from Baseline (week 2), at each of weeks 4,8,12,16,20, week 24 Final Study visit, and week 26 follow-up phone call. Will also be done for a study drug withdrawal visit or if applicable, an edaravone initiation visit.
  Adverse events will be assessed.
Change in ALS-Specific QOL -Revised | Change from Baseline (week 2), at week 24 Final Study visit. Will also be done for a study drug withdrawal visit or if applicable, an edaravone initiation visit.
  The Amyotrophic Lateral Sclerosis Specific Quality of Life - Revised (ALSSQOL-R) questionnaire consists of 50 items regarding quality of life. Takes approximately 15 minutes to complete
Change in Cramp Frequency and Severity | Change from Baseline (week 2), at each of weeks 4,8,12,16,20, and week 24 Final Study visit. Will also be done for a study drug withdrawal visit or if applicable, an edaravone initiation visit
  Consists of 2 questions asking if subject has had cramps in the last 24 hours, how bad and how severe they were. Takes 1 or 2 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Korngut, M.D., Principal Investigator — University of Calgary and Alberta Health Services
Locations (9):
- Canada (9):
  - Dr. Lawrence Korngut -South Health Campus, Calgary, Alberta
  - Dr. Wendy Johnston - University of Alberta, Edmonton, Alberta
  - Dr. Colleen O'Connell - Stan Cassidy Centre for Rehabilitation, Fredericton, New Brunswick
  - Dr. John Turnbull McMaster University/Hamilton Health Services, Hamilton, Ontario
  - Dr. Christen Shoesmith - London Health Sciences Centre, London, Ontario
  - Dr. Ariel Breiner -Ottawa Hospital Research Institute, Ottawa, Ontario
  - Dr. Lorne Zinman Sunnybrook Research Institute, Toronto, Ontario
  - Dr. Sandrine Larue - Reserche Sepmus Inc., Greenfield Park, Quebec
  - Dr. Genevieve Matte, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No